CLINICAL TRIAL: NCT01803204
Title: Evaluation of an Educational Booklet for Perioperative Orthognathic Surgery: Randomized Clinical Trial.
Brief Title: Patient Education Before Orthognathic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Cristina Silva Sousa, Student PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 193.454
Record Dates: First submitted 2013-02-25; First posted 2013-03-04 (Estimated); Results first posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2018-08

CONDITIONS: Malocclusion; Anxiety; Micrognathism; Prognathism
Keywords: Anxiety; Orthognathic surgery; Patient educational as topic; Patient educational handout; Pamphlets
MeSH Terms: conditions — Malocclusion; Anxiety Disorders; Micrognathism; Prognathism

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Booklet - Preoperative Educational (Experimental): This group received the booklet in the preoperative consult, they will monitoring during the postoperative phase
  Interventions: Other: Booklet - Preoperative Educational
- Control (No Intervention): This group don't received booklet, they will be monitored during the postoperative period to control

INTERVENTIONS:
Other: Booklet - Preoperative Educational — the patients receive a booklet during the preoperative phase. The educational session with a booklet will occur before the surgery.
  Arms: Booklet - Preoperative Educational

SUMMARY:
To evaluate the effectiveness in the use of an educational material through: Assessment of knowledge about post-operative orthognathic surgery; assessing levels of anxiety with the survey of Anxiety Inventory-STATE-TRAIT; clinical evaluation of self-care in the management of postoperative signs and symptoms

DETAILED DESCRIPTION:
It is a clinical randomized controlled trial being developed from February 2013 to September 2015, divided into two phases: a pilot study without randomization for impact testing and evaluation of intervention and, in the second time, the clinical randomized study with possible changes after the pilot study.

Will be entered in the study patients undergoing maxillofacial surgery originating at outpatient clinic located in the municipality of São Paulo. The study aims to evaluate the effects of educational material in postoperative education orthognathic surgery, with intervals between pre and postoperative serials.

Recruitment plan of patients: the patients seen in oral and maxillofacial surgery and traumatology clinic located in the municipality of São Paulo with indication for orthognathic surgery will be covered by personally and invited to participate in intervention research. To control the bias will be included in the study patients of the same surgical team, to ensure the same surgical technique and postoperative guidance conduct by the surgeon.

Study variables: it is intended to analyse the socio-demographic variables: sex, age, level of education; independent variables: surgical technique, recovery time, difficulties experienced during the postoperative period, possible surgical complications; dependent variables: signs and symptoms postoperatively (presence or absence) and monitoring of care during the postoperative period; level of knowledge about the post-op of orthognathic surgery and anxiety levels (State-trait anxiety inventory-IDATE).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing orthognathic surgery during the study and with surgical technique:

  * sagittal maxillary bilateral osteotomy;
  * maxillary;
  * vertical osteotomy;
  * Lefort I osteotomy combined with or without mentoplastia and maxillary disjunction.
* Informed consent
* Patients in the maxillofacial outpatient clinic located at Sao Paulo

Exclusion Criteria:

* patients undergoing reoperation of orthognathic surgery;
* with cleft lip-palate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina S Sousa, MsC, Principal Investigator — University of Sao Paulo
Locations (1):
- Cristina Silva Sousa, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] dos Santos MR, Sousa CS, Turrini RN. [Perception of orthognathic surgery patients on postoperative care]. Rev Esc Enferm USP. 2012 Oct;46 Spec No:78-85. doi: 10.1590/s0080-62342012000700012. Portuguese. PMID 23250262
- [Background] Sousa CS, Turrini RNT. Validação de constructo de tecnologia educativa para pacientes mediante aplicação da técnica Delphi. Acta Paulista de Enfermagem. 2012;25(6):990-6.
- [Background] Sousa CS, Turrini RN. Creating and validating educational material for patients undergoing orthognathic surgery. Asian Nurs Res (Korean Soc Nurs Sci). 2012 Dec;6(4):166-72. doi: 10.1016/j.anr.2012.10.006. Epub 2012 Nov 7. PMID 25031119
- [Background] Sousa CS, Turrini RNT. Complications in orthognathic surgery: A comprehensive review. Journal of Oral and Maxillofacial Surgery, Medicine, and Pathology. 2012;24:67-74.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For the pilot study and testing of the evaluation printed were contacted 8 patients as intervention group and control group not applied.
Period: Overall Study
Arm/Group | Booklet - Preoperative Educational | Control
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Booklet - Preoperative Educational | Control | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 3 | 5
  Between 18 and 65 years | 18 | 17 | 35
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (8.2) | 27.4 (6.9) | 27.1 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 11 | 9 | 20
Region of Enrollment [Number; unit: participants]
  Brazil | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Clinical Changes During the Postoperative Recovery
Description: A review of the patient's recovery after surgery will occur during follow-up visits with the surgeon, It was rated the care of oral hygiene, nutrition, mobility and sensitivity, appearance of lips, swelling, pain and sleep . The patient will be accompanied by the researcher during the return and the data will be evaluated and investigated as annotated patient outcomes.
Time Frame: this measure will be assessed weekly in the first forty days postoperatively (seventh day, fourteenth day, twenty-first day and fortieth day after the surgery)
Measure: Number; unit: participants
Arm/Group | Booklet - Preoperative Educational | Control
Number analyzed (Participants) | 20 | 20
participants | 10 | 10
Statistical Analysis 1: Comparison: Booklet - Preoperative Educational vs Control; Test type: Superiority or Other; p = 1.00, GEE; GEE = 1.00

2. Secondary Outcome: Average Test Arrangements on Surgery
Description: The patient's knowledge about the surgery will be assessed by a test developed by the researcher (A test with 10 multiple choice questions, each questions with 4 alternatives, about care after surgery. Each questions value 1 point, for better results was considered higher 7 points and for worse results was considered low 5 points. A total value for the Knowledge test was 10 points (rage 0-10) The acceptable score to understand that the patient is aware of the surgery was 7.
  This was applied on two occasions: first contact with the patient before surgery, signed a consent form before the start researcher educational intervention (during the preoperative phase).
  The second test will be given at the first follow-up visit with the surgeon (seventh postoperative day)
Time Frame: This will be delivered in the first contact with the patient before surgery and on the seventh day after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Booklet - Preoperative Educational | Control
Number analyzed (Participants) | 20 | 20
score on a scale
  Pos-op First visit | 6.5 (1.53) | 4.3 (1.94)
  Pos -op Thrid visit | 6.8 (1.64) | 5.0 (2.21)
  Pos-op Fourth visit | 7.00 (1.55) | 5.20 (2.32)
  Pre-operatively | 4.20 (1.72) | 4.30 (2.22)
Statistical Analysis 1: Comparison: Booklet - Preoperative Educational vs Control; Test type: Superiority or Other; p < 0.01, Mist Effects Model

3. Other Pre Specified Outcome: Levels of Anxiety After Educational Intervention
Description: The levels of anxiety during the perioperative period will be measured with the State-Trait Anxiety Inventory (STAI).
  The STAI has 40 items, 20 items allocated to each of the S-Anxiety and T-Anxiety sub-scales Responses for the S-Anxiety scale assess intensity of current feelings "at this moment": 1) not at all, 2) somewhat, 3) moderately so, and 4) very much so. Responses for the T-Anxiety scale assess fre- quency of feelings "in general": 1) almost never, 2) some- times, 3) often, and 4) almost always.
  Scoring. Item scores are added to obtain subtest total scores. Scoring should be reversed for anxiety-absent items (19 items of the total 40).
  Score interpretation. Range of scores for each subtest is 20-80, the higher score indicating greater anxiety. A cut point of 39-40 has been suggested to detect clinically significant symptoms for the S-Anxiety scale For results this intervention was considered S-STAI Anxiety with lower scores (< 39) after the intervention
Time Frame: The STAI will be applied on the seventh day after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Booklet - Preoperative Educational | Control
Number analyzed (Participants) | 20 | 20
score on a scale
  Pre-operatively S-STAI anxiety | 39.30 (12.13) | 45.20 (10.45)
  Pos -op First visit S-STAI anxiety | 35.8 (11.37) | 40.10 (11.24)
  Pos-op Third visit S-STAI anxiety | 33.90 (9.41) | 36.70 (10.39)
  Pos-op Fourth visit S-STAI anxiety | 34.40 (10.21) | 37.20 (10.46)
Statistical Analysis 1: Comparison: Booklet - Preoperative Educational vs Control; Test type: Superiority or Other; p = 0.81, Mist Effect Model

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Booklet - Preoperative Educational | Control
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
It's possible lack of patient adherence to educational intervention, which would lead to lower intervention response rates and the possible use of other technologies during the process.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No